CLINICAL TRIAL: NCT03057600
Title: A Multicenter Phase 2 Study of the Glutaminase Inhibitor CB-839 in Combination With Paclitaxel in Patients With Advanced Triple Negative Breast Cancer (TNBC) Including Patients of African Ancestry and Non-African Ancestry
Brief Title: Study of CB-839 in Combination w/ Paclitaxel in Participants of African Ancestry and Non-African Ancestry With Advanced Triple Negative Breast Cancer (TNBC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX-839-007
Record Dates: First submitted 2017-02-10; First posted 2017-02-20 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Triple Negative Breast Cancer; TNBC - Triple-Negative Breast Cancer
Keywords: African ancestry; African American; CB-839; Glutaminase Inhibitor; Glutaminase; TNBC; Tumor Metabolism; Glutamine
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Paclitaxel; taxane; CB-839

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of 4 arms depending on the number of prior lines of therapy they have received and whether or not they have African ancestry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - African ancestry, 3rd line+ (Experimental): Intervention = Paclitaxel- CB-839 (Pac-CB) combination
  1. Participants must self-identify as African ancestry (includes African American).
  2. At least 2 prior lines of systemic therapy for advanced/metastatic disease including a taxane.
     * Prior taxane (paclitaxel, docetaxel, or nab-paclitaxel) for advanced/metastatic disease is required but must not have been received in the immediate prior line of therapy.
     * Systemic neoadjuvant and/or adjuvant therapy is considered a line of therapy for advanced/metastatic disease if the time to recurrence from completion of treatment was ≤ 12 mo.
  Interventions: Drug: Paclitaxel; Drug: CB-839
- Cohort 2 - African ancestry, 1st line (Experimental): Intervention = Pac-CB combination
  1. Participants must self-identify as African ancestry (includes African American).
  2. No prior systemic therapy for advanced or metastatic disease.
     * Systemic neoadjuvant or adjuvant therapy, including taxane, is allowed if time to recurrence was > 12 mo.
  Interventions: Drug: Paclitaxel; Drug: CB-839
- Cohort 3 - Non-African ancestry, 3rd line+ (Experimental): Intervention = Pac-CB combination
  1. Participants do not self-identify as African ancestry.
  2. Otherwise have the same criteria as Cohort 1.
  Interventions: Drug: Paclitaxel; Drug: CB-839
- Cohort 4 - Non-African ancestry, 1st line (Experimental): Intervention = Pac-CB combination
  1. Participants do not self-identify as African ancestry.
  2. Otherwise have the same criteria as Cohort 2.
  Interventions: Drug: Paclitaxel; Drug: CB-839

INTERVENTIONS:
Drug: Paclitaxel — standard weekly paclitaxel in 28-day cycles
  Other Names: Taxane
Drug: CB-839 — CB-839 administered as oral tablets twice daily (BID)
  Other Names: telaglenastat

SUMMARY:
CX-839-007 is an open-label Phase 2 study of the combination of CB-839 with paclitaxel in participants of African ancestry and non-African ancestry with advanced triple negative breast cancer. Multiple single-arm cohorts will be enrolled in which 800 mg twice daily (BID) CB-839 will be administered in combination with the full approved dose of paclitaxel.

DETAILED DESCRIPTION:
Participants will be enrolled into 4 cohorts, as follows:

* Cohort 1: patients of African ancestry with 2 or more lines of prior therapy for metastatic disease
* Cohort 2: patients of African ancestry with no prior lines of therapy for metastatic disease
* Cohort 3: same as cohort 1 but in patients of non-African ancestry
* Cohort 4: same as cohort 2 but in patients of non-African ancestry

ELIGIBILITY:
Key Inclusion Criteria:

* Meets criteria for 1 of the 4 defined study cohorts
* TNBC, defined as estrogen receptor (ER) and progesterone receptor (PR) negative (< 1% by immunohistochemistry) and human epidermal growth factor receptor 2 (HER2)-negative (immunohistochemistry 0 to 1+ or fluorescence in situ hybridization [FISH] negative)
* Metastatic disease or locally-advanced disease not amenable to curative intent treatment
* Adequate hepatic, renal, cardiac, and hematologic function
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Recovery to baseline or ≤ Grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version.4.0

Key Exclusion Criteria:

* Known brain metastases or central nervous system (CNS) cancer unless adequately treated with radiotherapy and/or surgery and stable for ≥ 2 mo
* Unable to receive oral medications
* Known hypersensitivity to Cremophor®-based agents
* Major surgery within 28 days of Cycle 1 Day 1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Whiting, MD, PhD, Study Director — Calithera Biosciences, Inc
Locations (25):
- United States (25):
  - University of Alabama at Brimingham, Birmingham, Alabama
  - University of South Alabama, Mitchell Cancer Institute, Mobile, Alabama
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University Cancer and Blood Center, Athens, Georgia
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - Northwest Georgia Oncology, Marietta, Georgia
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Louis University, St Louis, Missouri
  - JTCC at Hackensack UMC, Hackensack, New Jersey
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Womens Hospital - UPMC, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Greenville Health System (GHS) Cancer Institute, Greenville, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson, Houston, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - African Ancestry, 3rd Line+: Participants self-identifying as African ancestry (includes African American) with at least 2 prior lines of systemic therapy for advanced/metastatic disease including a taxane, received 800 mg CB-839 tablets orally (PO) twice daily (BID) on Days 1 through 28 of each 28-day cycle along with 80 mg/m^2 of paclitaxel intravenous (IV) infusion on Days 1, 8, and 15 of each 28-day cycle until disease progression, unacceptable toxicity, initiation of another systemic anticancer treatment, death, or withdrawal of consent.
- Cohort 2 - African Ancestry, 1st Line: Participants self-identifying as African ancestry (includes African American) with no prior systemic therapy for advanced or metastatic disease received 800 mg CB-839 tablets PO BID on Days 1 through 28 of each 28-day cycle along with 80 mg/m^2 of paclitaxel IV infusion on Days 1, 8, and 15 of each 28-day cycle until disease progression, unacceptable toxicity, initiation of another systemic anticancer treatment, death, or withdrawal of consent.
- Cohort 3 - Non-African Ancestry, 3rd Line+: Participants not self-identifying as African ancestry (includes African American) with at least 2 prior lines of systemic therapy for advanced/metastatic disease including a taxane, received 800 mg CB-839 tablets PO BID on Days 1 through 28 of each 28-day cycle along with 80 mg/m^2 of paclitaxel IV infusion on Days 1, 8, and 15 of each 28-day cycle until disease progression, unacceptable toxicity, initiation of another systemic anticancer treatment, death, or withdrawal of consent.
- Cohort 4 - Non-African Ancestry, 1st Line: Participants not self-identifying as African ancestry (includes African American) with no prior systemic therapy for advanced or metastatic disease received 800 mg CB-839 tablets PO BID on Days 1 through 28 of each 28-day cycle along with 80 mg/m^2 of paclitaxel IV infusion on Days 1, 8, and 15 of each 28-day cycle until disease progression, unacceptable toxicity, initiation of another systemic anticancer treatment, death, or withdrawal of consent.
Period: Overall Study
Arm/Group | Cohort 1 - African Ancestry, 3rd Line+ | Cohort 2 - African Ancestry, 1st Line | Cohort 3 - Non-African Ancestry, 3rd Line+ | Cohort 4 - Non-African Ancestry, 1st Line
Started | 9 | 10 | 20 | 13
Completed | 0 | 0 | 0 | 0
Not Completed | 9 | 10 | 20 | 13
Not completed — Adverse Event | 0 | 0 | 4 | 0
Not completed — Radiologic Disease Progression | 8 | 7 | 13 | 10
Not completed — Symptomatic Deterioration | 0 | 1 | 1 | 0
Not completed — Investigator Decision | 0 | 0 | 1 | 0
Not completed — Study Termination by Sponsor | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Other, Not Specified | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - African Ancestry, 3rd Line+ | Cohort 2 - African Ancestry, 1st Line | Cohort 3 - Non-African Ancestry, 3rd Line+ | Cohort 4 - Non-African Ancestry, 1st Line | Total
Number analyzed (Participants) | 9 | 10 | 20 | 13 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (9.40) | 64.0 (8.68) | 55.8 (13.02) | 59.5 (11.13) | 57.3 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 20 | 13 | 52
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 0 | 3
  Not Hispanic or Latino | 9 | 10 | 17 | 13 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 9 | 10 | 0 | 0 | 19
  White | 0 | 0 | 17 | 13 | 30
  Other, Not Specified | 0 | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of patients with complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1criteria:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessment performed no less than 4 weeks after the criteria for response were first met.
Time Frame: Maximum duration of follow-up for ORR was 14.8 months.
Population: Response Evaluable Analysis Set: all participants who had measurable disease at baseline, received at least 1 dose of study drug (telaglenastat or paclitaxel) and completed at least 1 post baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 - African Ancestry, 3rd Line+ | Cohort 2 - African Ancestry, 1st Line | Cohort 3 - Non-African Ancestry, 3rd Line+ | Cohort 4 - Non-African Ancestry, 1st Line
Number analyzed (Participants) | 9 | 10 | 19 | 13
percentage of participants | 22.2 [2.8 to 60.0] | 10.0 [0.3 to 44.5] | 10.5 [1.3 to 33.1] | 53.8 [25.1 to 80.8]
Statistical Analysis 1: Comparison: Cohort 1 - African Ancestry, 3rd Line+; Test type: Superiority; p = 0.2252, exact one-sample binomial tests
Statistical Analysis 2: Comparison: Cohort 2 - African Ancestry, 1st Line; Test type: Superiority; p = 0.9437, exact one-sample binomial tests
Statistical Analysis 3: Comparison: Cohort 3 - Non-African Ancestry, 3rd Line+; Test type: Superiority; p = 0.5797, exact one-sample binomial tests
Statistical Analysis 4: Comparison: Cohort 4 - Non-African Ancestry, 1st Line; Test type: Superiority; p = 0.0243, exact one-sample binomial tests

2. Secondary Outcome: Progression Free Survival (PFS) as Assessed by Investigator
Description: PFS was defined as time from the first dose date to the earlier of either progression of disease per RECIST v1.1 or death from any cause. The duration of progression-free survival was censored at the date of last radiographic disease if the patient was alive and progression free at the time of analysis data cutoff, disease progression or death occurred after missing data for 2 consecutive radiographic disease assessments, or patient received non-protocol TNBC treatment prior to documentation of disease progression. Kaplan-Meier product-limit estimates. Brookmeyer-Crowley methodology for a non-parametric 95% confidence interval (CI) is used.
  Progressive Disease (PD) per RECIST 1.1: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Maximum duration of follow-up for PFS was 17.0 months.
Population: PFS Evaluable Analysis Set: all participants who received at least 1 dose of any study-specific treatment (telaglenastat or paclitaxel).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohort 1 - African Ancestry, 3rd Line+: Participants self-identifying as African ancestry (includes African American) with at least 2 prior lines of systemic therapy for advanced/metastatic disease including a taxane, received 800 mg CB-839 tablets PO BID on Days 1 through 28 of each 28-day cycle along with 80 mg/m^2 of paclitaxel IV infusion on Days 1, 8, and 15 of each 28-day cycle until disease progression, unacceptable toxicity, initiation of another systemic anticancer treatment, death, or withdrawal of consent.
Arm/Group | Cohort 1 - African Ancestry, 3rd Line+ | Cohort 2 - African Ancestry, 1st Line | Cohort 3 - Non-African Ancestry, 3rd Line+ | Cohort 4 - Non-African Ancestry, 1st Line
Number analyzed (Participants) | 9 | 10 | 20 | 13
months | 2.30 [1.74 to 3.48] | 5.49 [1.84 to 5.72] | 2.00 [1.64 to 3.38] | 7.33 [3.71 to 16.46]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the first dose date to death due to any cause. For patients alive at time of analysis, overall survival will be censored at the time when the patient is last known to be alive.Kaplan-Meier product-limit estimates. Brookmeyer-Crowley methodology for a non-parametric 95% CI is used. Median is defined to be the smallest observed survival time for which the value of the estimated survival function is less than or equal to 0.5.
Time Frame: Maximum duration of follow-up for OS was 24.1 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 - African Ancestry, 3rd Line+ | Cohort 2 - African Ancestry, 1st Line | Cohort 3 - Non-African Ancestry, 3rd Line+ | Cohort 4 - Non-African Ancestry, 1st Line
Number analyzed (Participants) | 9 | 10 | 20 | 13
months | 7.26 [5.09 to 16.95] | 13.47 [6.97 to 14.69] | 6.44 [2.73 to 8.84] | 16.76 [12.88 to NA] — Not estimable due to small number of events.

4. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is defined as the time between the first documentation of a confirmed PR or a CR to the first documentation of PD or death, whichever occurs first. The duration of response will be censored at the date of last radiographic disease if the patient is alive and progression free at the time of database lock, disease progression or death occurs after missing data for two consecutive radiographic disease assessments, or patient receives non-protocol TNBC treatment prior to documentation of disease progression.
  RECIST v1.1 criteria:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Maximum duration of follow-up for DOR was 14.8 months.
Population: Response Evaluable Analysis Set: all participants who had measurable disease at baseline, received at least 1 dose of study drug (telaglenastat or paclitaxel) and completed at least 1 post baseline tumor assessment. Participants defined as responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 - African Ancestry, 3rd Line+ | Cohort 2 - African Ancestry, 1st Line | Cohort 3 - Non-African Ancestry, 3rd Line+ | Cohort 4 - Non-African Ancestry, 1st Line
Number analyzed (Participants) | 2 | 1 | 2 | 7
months | NA [3.68 to NA] — Not Estimable. Among the 2 participants analyzed, 1 participant was censored for duration of response. Median and upper bound of 95% confidence interval could not be estimated based on uncensored data from 1 participant. | 6.47 [NA to NA] — 95% confidence interval not calculable because data were only collected for 1 participant. | 7.61 [4.07 to 11.14] | 11.04 [5.55 to 14.75]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate is defined as the percentage of patients with best response of CR, PR, or SD per RECIST v1.1 criteria lasting ≥ 16 weeks for 3rd line + patients and ≥ 24 weeks for 1st line patients. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Maximum duration of follow-up for CBR was 14.8 months.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 - African Ancestry, 3rd Line+ | Cohort 2 - African Ancestry, 1st Line | Cohort 3 - Non-African Ancestry, 3rd Line+ | Cohort 4 - Non-African Ancestry, 1st Line
Number analyzed (Participants) | 9 | 10 | 19 | 13
percentage of participants | 22.2 [2.8 to 60.0] | 20.0 [2.5 to 55.6] | 10.5 [1.3 to 33.1] | 61.5 [31.6 to 86.1]

ADVERSE EVENTS:
Time Frame: All Cause Mortality: from enrollment through study follow-up. Maximum duration of follow-up was 24.1 months. Adverse Events: from first dose of study drug through end of treatment (EOT) + 28 days post treatment discontinuation. Median duration of treatment was 84 days for COhort 1, 118 days for Cohort 2, 51.0 days for Cohort 3, and 224.0 days for Cohort 4.
Description: Per protocol, Grade 5 disease progression events are excluded from these tables. Disease progression includes events in the preferred terms of disease progression and malignant neoplasm progression.
Arm/Group | Cohort 1 - African Ancestry, 3rd Line+ | Cohort 2 - African Ancestry, 1st Line | Cohort 3 - Non-African Ancestry, 3rd Line+ | Cohort 4 - Non-African Ancestry, 1st Line
All-Cause Mortality (participants affected / at risk) | 7/9 | 7/10 | 14/20 | 7/13
Serious Adverse Events (participants affected / at risk) | 2/9 | 2/10 | 5/20 | 2/13
Other Adverse Events (participants affected / at risk) | 9/9 | 10/10 | 19/20 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - African Ancestry, 3rd Line+ (N=9) | Cohort 2 - African Ancestry, 1st Line (N=10) | Cohort 3 - Non-African Ancestry, 3rd Line+ (N=20) | Cohort 4 - Non-African Ancestry, 1st Line (N=13)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - African Ancestry, 3rd Line+ (N=9) | Cohort 2 - African Ancestry, 1st Line (N=10) | Cohort 3 - Non-African Ancestry, 3rd Line+ (N=20) | Cohort 4 - Non-African Ancestry, 1st Line (N=13)
Fatigue (General disorders) | 5 | 3 | 10 | 10
Oedema peripheral (General disorders) | 0 | 2 | 3 | 4
Chest pain (General disorders) | 2 | 0 | 2 | 1
Pyrexia (General disorders) | 1 | 0 | 3 | 1
Pain (General disorders) | 0 | 0 | 2 | 2
Chills (General disorders) | 0 | 0 | 0 | 3
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 2 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0
Axillary pain (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1 | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 5 | 4
Constipation (Gastrointestinal disorders) | 2 | 2 | 3 | 5
Vomiting (Gastrointestinal disorders) | 1 | 1 | 5 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral herpes (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 4 | 1 | 2 | 5
Dizziness (Nervous system disorders) | 2 | 1 | 6 | 0
Headache (Nervous system disorders) | 1 | 2 | 2 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 2 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Jugular vein occlusion (Nervous system disorders) | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 4 | 7 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 6 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4 | 5 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 4 | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 3 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 3 | 5
White blood cell count decreased (Investigations) | 2 | 3 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 3 | 3
Neutrophil count decreased (Investigations) | 1 | 1 | 3 | 2
Weight decreased (Investigations) | 1 | 1 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 1
Platelet count decreased (Investigations) | 1 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Nail bed disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pustular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Scratch (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 5 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 3
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Bacterial vaginosis (Infections and infestations) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 2 | 0 | 4 | 1
Vision blurred (Eye disorders) | 1 | 0 | 1 | 2
Vitreous floaters (Eye disorders) | 1 | 2 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 2
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 3 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Recall phenomenon (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication by the PI before either a multi-site publication or 18 months after final multi-site study report. PI can only publish their own results and provide 45 days in advance notice. PI must delete any Calithera confidential information from the publication other than study results and give good faith consideration to other comments made by Calithera. The PI must delay the publication for up to 45 days if requested by Calithera and publicly acknowledge Calithera and Pfizer support.

DOCUMENTS (2):
  • Study Protocol (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03057600/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03057600/SAP_001.pdf